CLINICAL TRIAL: NCT07271901
Title: Masticatory Performance in Mixed Dentition Children Before and After Dental Treatment: an in Vivo Assessment Using a Two-coloured Chewing Gum Mixing Test
Brief Title: Masticatory Performance in Mixed Dentition Children Before and After Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ezgi Turkyilmaz, Research Assistant, Department of Pediatric Dentistry, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERU-PEDO-2025-MP01
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Dental Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental Treatment (Experimental)
  Interventions: Other: Dental Treatment

INTERVENTIONS:
Other: Dental Treatment — Comprehensive dental treatment including restorative procedures, pulp therapy, and extractions performed under local anesthesia as indicated. The intervention aimed to eliminate dental caries and restore normal oral function. Masticatory performance was evaluated before and three months after treatment using a two-coloured chewing gum mixing test and analyzed with ViewGum© software to assess improvement in chewing ability.

SUMMARY:
This prospective clinical study aimed to evaluate the effects of dental treatment on masticatory performance and food preferences in children during the mixed dentition period. A total of 100 children aged 6 to 9 years were included and categorized into three groups based on the Caries Assessment Spectrum and Treatment (CAST) index (CAST 5, 6, and 7). Masticatory performance was objectively assessed using a two-coloured chewing gum mixing test (Vivident Fruit Swing) and analyzed with ViewGum© software by calculating the Variance of Hue (VOH) value. Assessments were performed before and three months after dental treatment. Additional variables such as posterior occlusal contacts, body mass index (BMI), and pain scores were also recorded. The study aimed to determine the improvement in masticatory function and the potential association between oral rehabilitation and food preference changes in children during the mixed dentition period.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 9 years in the mixed dentition period Presence of dental caries categorized as CAST codes 5, 6, or 7 Children with fully erupted permanent first molars Medically healthy children (ASA I) Cooperative or manageable with nonpharmacological behavior guidance techniques Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Children with systemic or neurological disorders affecting mastication or swallowing History of orthodontic or prosthetic treatment Presence of temporomandibular joint dysfunction Use of medications influencing salivary flow or muscle activity Uncooperative children for whom the chewing test could not be standardized

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Variance of Hue (VOH) Values Before and After Dental Treatment | Baseline and 3 months after dental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Turkyilmaz, Principal Investigator — Erciyes University Faculty of Dentistry
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No